CLINICAL TRIAL: NCT05516992
Title: A Phase 3, Multi-center, Randomized, Double-blind, Placebo-controlled Study, to Evaluate the Safety and Efficacy of SB-01 For Injection for the Treatment of Lumbar Degenerative Disc Disease
Brief Title: Moderate - Severe Degenerative Disc Disease Evaluation of the Lumbar Spine
Acronym: MODEL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Spine BioPharma, Inc (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SB01-M001
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, placebo-controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SB-01 For Injection (Experimental): Subjects receive a SB-01 For Injection intradiscal injection per treated disc.
  Interventions: Drug: SB-01 For Injection
- Sham Needle (Placebo Comparator): Subjects receive a sham needle placement for each treated disc.
  Interventions: Drug: Sham Needle

INTERVENTIONS:
Drug: SB-01 For Injection — Intradiscal injection
  Arms: SB-01 For Injection
Drug: Sham Needle — Sham needle placement
  Arms: Sham Needle

SUMMARY:
The purpose of the study is to confirm the safety and effectiveness of SB-01 For Injection in adult patients with chronic low back pain and related disability due to Lumbar Degenerative Disc Disease. The primary effectiveness hypothesis is superiority of the investigational product relative to control in terms of the percentage of subjects improving in pain-related disability.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Back pain greater than 'worst leg pain' as measured by the NRS
3. Diagnosed with one or two contiguous level(s) lumbar (L1-S1) disc degeneration of Pfirrmann Grade 3 and/or 4 determined by MRI analyzed by the independent radiologic central lab
4. Have chronic low back pain and related disability for at least 6 months with at least 3 months of prior conservative treatment
5. Baseline ODI score ≥ 40/100
6. Baseline NRS ≥ 4 points (Back)
7. Willing and able to provide Informed Consent for study participation
8. Willing and able to comply with this protocol and be available for the entire duration of the study, including ability to access the internet
9. Must practice effective contraception during the first 3 months of follow-up (female of childbearing potential and male subjects):

   1. Abstinence or,
   2. Surgical Sterilization or,
   3. Oral Contraceptives or,
   4. Barrier Methods (Condoms, IUD's).
10. Patient must verify that:

    1. In the case of females, the patient is post-menopausal or is surgically sterile or,
    2. In the case of males, the patient is surgically sterile or,
    3. The patient (male or female) confirms that they are at a point in their life where they are beyond consideration of having children.

Exclusion Criteria:

To qualify for enrollment in this study, patients must meet none of the exclusion criteria as follows.

1. Prior epidural, sacroiliac joint, and facet injections, or facet RFA (radiofrequency ablations) at any lumbosacral level within the past 4 weeks (e.g., transforaminal, interlaminar, caudal)
2. Prior interventional procedures of other types at any lumbosacral level at any time (e.g., intradiscal injection, basivertebral nerve ablation, biacuplasty, spinal cord stimulator, others)
3. Prior spine surgery at any lumbosacral level at any time (e.g., discectomy, decompression, instrumentation, fusion, fracture treatment, others)
4. Prior fracture at any lumbar level
5. Significant neurologic symptoms:

   1. Grade 3/5 or lower strength in any lumbar myotome
   2. Sensory deficit in a clearly radicular or sensory dermatome
6. MRI evidence of disc height loss > 2/3 of adjacent disc at any level to be injected, determined by the independent radiologic central lab
7. MRI evidence of other disc degeneration: Pfirrmann Grade 3-5 at any level not to be injected, determined by the independent radiologic central lab
8. MRI evidence of disc herniation with neural compression at any level, determined by the independent radiologic central lab
9. MRI evidence of significant stenosis of the central canal at any level, determined by the independent radiologic central lab
10. MRI evidence of foraminal stenosis with neural compression at any level, determined by the independent radiologic central lab
11. MRI evidence of moderate-to-severe facet arthrosis with edema at any level, determined by the independent radiologic central lab
12. Spondylolisthesis (antero or retrolisthesis) > 25% at any level, determined by the independent radiologic central lab
13. Lumbar coronal deformity, determined by the independent radiologic central lab:

    a. L1-S1 regional deformity > 25 degrees
14. Spondylolysis at any level
15. Lumbar inflammatory spondylitis
16. Recent history (previous six months) of chemical or alcohol dependence
17. Chronic narcotic use for more than defined as a daily dose of greater than 40 Morphine Equivalent Units (MEUs)
18. Depression or Somatization defined through the Distress and Risk Assessment Method (DRAM) scoring with Zung score > 33 or Zung > 17 and the Modified Somatic Perception Questionnaire (MSPQ) score > 12
19. Extreme obesity, defined by NIH Clinical Guidelines Body Mass Index (BMI > 40)
20. A QT duration corrected for heart rate by Fridericia's formula (QTcF) > 470 millisecond (msec)
21. Active systemic infection
22. Infection at the site of procedure pre-operatively
23. Cauda equina syndrome or neurogenic bowel/bladder dysfunction
24. Any terminal, systemic, or autoimmune disease including fibromyalgia, which may, in the opinion of the Principal Investigator compromise a subject's ability to comply with study procedures, and/or confound data
25. Metabolic bone disease (e.g., osteoporosis/osteopenia, gout, osteomalacia, Paget's disease)
26. Any disease, condition or surgery which might impair healing, such as:

    1. Active malignancy
    2. History of metastatic malignancy
27. Currently experiencing an episode of major mental illness (psychosis, major affective disorder, or schizophrenia), or manifesting physical symptoms without a diagnosable medical condition to account for the symptoms, which may indicate symptoms of psychological rather than physical origin
28. Any planned surgical procedure within the subject participation period (screening through the 12 Month Visit)
29. Any clinically relevant laboratory result on the screening visit Chem-12, hematology, or coagulation panels
30. Pregnancy at the time of screening, randomization, or planning to become pregnant during the first 3 months of follow-up
31. Currently a prisoner
32. Participation in any other investigational drug, biologic, or medical device study within the last 6 months prior to study procedure
33. Receiving Work Compensation benefits or engaged in personal spinal injury medical/legal litigation
34. Patient cannot be currently using the prohibited medications listed in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-08-27 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in function on the Oswestry Disability Index (ODI) at 6 months. | Baseline/Screening and 6 Month
  The ODI is a validated, 10-item self-reported instrument assessment of pain-related disability. Possible scores range from 0 (no disability) - 50 (severe disability). Further calculations are applied to reach a percentage score.

SECONDARY OUTCOMES:
Change from Baseline in pain on the Numerical Rating Scale (NRS) at 6 months. This outcome will only be tested if the primary endpoint is met. | Baseline/Screening and 6 Month
  The NRS is an 11-point scale, self-reported instrument assessment of pain intensity ranging across a continuum from no pain to an extreme amount of pain. The NRS will be collected for: Back and both legs. A lower score indicates less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gilligan, MD, MBA, Principal Investigator — Brigham and Women's Spine Center
Locations (29):
- United States (29):
  - Central Alabama Research, Birmingham, Alabama
  - Evolve Clinical Research, Phoenix, Arizona
  - Neurovations Research, Napa, California
  - Source Healthcare, Santa Monica, California
  - Science Connections, LLC, Doral, Florida
  - Coastal Clinical Research, Jacksonville, Florida
  - Conquest Research, Orlando, Florida
  - Pain Relief Centers, St. Petersburg, Florida
  - Tampa Pain Relief Center, Tampa, Florida
  - Florida Pain Relief Group, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Vista Clinical Research, LLC, Newnan, Georgia
  - Injury Care Research, Boise, Idaho
  - The Orthopaedic Research Foundation, Inc (OrthoIndy), Indianapolis, Indiana
  - Abay Neuroscience Center, Wichita, Kansas
  - OrthoNebraska, Omaha, Nebraska
  - Pioneer Clinical Research, New York, New York
  - Meta Medical Research Institute, Cincinnati, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - The Orthopedic Center, Tulsa, Oklahoma
  - HD Research, Bellaire, Texas
  - NeuroCare Partners, Houston, Texas
  - South Texas Spinal Clinic, San Antonio, Texas
  - Precision Spine Care, Tyler, Texas
  - Tranquil Clinical Research, Webster, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - Virginia iSpine Physicians, Richmond, Virginia
  - Gershon Pain Specialists, Virginia Beach, Virginia